CLINICAL TRIAL: NCT05923463
Title: A Scalable Service to Improve Health Care Quality Through Precision Audit and Feedback: A Cluster-randomized Controlled Trial
Brief Title: Precision Feedback to Improve Health Care Quality
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Library of Medicine (NLM) (NIH)
Responsible Party: Principal Investigator, Zach Landis-Lewis, Assistant Professor of Learning Health Sciences, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00194224; R01LM013894-01 (NIH)
Record Dates: First submitted 2023-06-20; First posted 2023-06-28 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Anesthesia Care Quality
Keywords: Audit and feedback; Anesthesiology; Learning health system

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- precision-enhanced feedback email messages (Experimental): Providers receive an enhanced monthly email containing precision audit and feedback (A&F).
  Interventions: Behavioral: precision-enhanced feedback email messages
- standard feedback email messages (Active Comparator): Providers receive the standard "one size fits most" A&F monthly email.
  Interventions: Behavioral: standard feedback email messages

INTERVENTIONS:
Behavioral: precision-enhanced feedback email messages — Providers receive customized messages prioritizing metrics in an optimal formatting.
  Arms: precision-enhanced feedback email messages
Behavioral: standard feedback email messages — Providers receive metrics in a common format.
  Arms: standard feedback email messages

SUMMARY:
This cluster-randomized trial will assess the effectiveness of a precision feedback service on anesthesia provider performance. The precision feedback service enhances a standard audit and feedback (A&F) email with a brief message and visual display about high-value performance information. The control arm will receive a standard "one size fits most" A&F email that is currently sent to anesthesia providers each month. Hypothesis: Providers receiving precision feedback will increase a) care quality for improvable measures and b) email engagement (click-through and dashboard login rates) when compared with providers receiving standard A&F emails. The study investigators will assess unintended consequences in a mixed-methods process evaluation.

ELIGIBILITY:
Inclusion Criteria (assessed before interventional period):

* Participation in the Multicenter Perioperative Outcomes Group (MPOG) provider feedback email program.

Exclusion Criteria (assessed after interventional period):

* Ended participation in the MPOG provider feedback email program for any reason during the study period
* Changed professional roles (e.g. transitioned from resident to attending) before the end of the intervention period
* Changed institutions during the study period
* Had no institution-selected quality measures in common between the pre-intervention and intervention period
* Were not candidates to receive a precision feedback email for the majority of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3500 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Measure success rate (M) for operative cases of anesthesia care providers | Up to 1 year
  The primary outcome for the cluster-randomized controlled trial is the measure success rate (M) for operative cases of anesthesia care providers, where:
  M = sum of all operative case measurement successes / number of all operative case measurements
  The measures included in each provider's measure success rate will be all improvable process measures that meet the following inclusion criteria:
  1. A provider's cases were included for the measure during both the 6-month pre-intervention period and during the 6-month intervention period.
  2. Average performance for the measure is below 90% during the baseline period, based on the MPOG threshold for most process measures.
  3. The measure was included in at least one provider feedback email during the intervention period.
  The investigators will exclude measures of clinical outcomes (also called "inverse measures") in this study that are less within the control of providers.

SECONDARY OUTCOMES:
Average email click-through rate (CTR) | Up to 6 months
  CTR = 100 x (number of recipient's emails with a clicked link) / (total number of emails)
Average dashboard login rate (L) | Up to 1 year
  L = 100 x (number of months with an email recipient's dashboard login event) / (total number of months)

CONTACTS AND LOCATIONS:
Overall Officials: Zach Landis-Lewis, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Landis-Lewis Z, Flynn A, Janda A, Shah N. A Scalable Service to Improve Health Care Quality Through Precision Audit and Feedback: Proposal for a Randomized Controlled Trial. JMIR Res Protoc. 2022 May 10;11(5):e34990. doi: 10.2196/34990. PMID 35536637